CLINICAL TRIAL: NCT01052415
Title: POL and Access Intervention to Reduce HIV Stigma Among Service Providers in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH081778 (NIH)
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: HIV-related Stigma; Patient Satisfaction; Provider-patient Interaction
Keywords: HIV; Stigma; POL; Service providers; China; Universal precaution
MeSH Terms: conditions — Patient Satisfaction; Social Stigma | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): Service providers and HIV patients, offered intervention at the end of study
- Intervention (Experimental): Behavioral: Cognitive-behavioral, small group format sessions delivered in Chinese to service providers and HIV patients.
  Interventions: Behavioral: Cognitive behavioral sessions

INTERVENTIONS:
Behavioral: Cognitive behavioral sessions — Behavioral: Cognitive-behavioral, small group format sessions delivered in Chinese to service providers and HIV patients.
  Other Names: Intervention, service providers, HIV-related stigma
  Arms: Intervention

SUMMARY:
In this project, UCLA's Center for Community Health (CCH) will develop an efficacious intervention trial integrating both individual and structural components to reduce HIV- related stigma among service providers in China and therefore benefit people living with HIV/AIDS (PLWHA).

The purpose of this study is to develop a feasible, practical and low cost intervention strategy that will prevent and/or reduce the negative effects of HIV-related stigma among health service providers in China.

This project will be conducted in two provinces and proceed in two phases. In Phase 1, confidential focus groups will take place with small samples of service providers and hospital administrators to finalize the intervention activities, and the investigators will also test and finalize the Audio Computer-Assisted Self-Interview (ACASI) assessment measures and implementation procedures with the same group of service providers. During Phase 1 a small sample of patients will anonymously test the paper-pencil baseline survey. Equal number of samples will be selected from two counties of each province. The findings from Phase 1 will be used to develop intervention, and revise assessment for Phase 2.

DETAILED DESCRIPTION:
HIV is a serious problem and HIV-related stigma in the medical setting is impeding every step in the battle against HIV in China. The number of annual reported HIV infections in China has increased steadily. The proposed study will be the first randomized controlled intervention trial that specifically targets stigma and access to universal precautions in medical settings, and is implemented at multiple sites in Yunnan and Fujian. Among the two target provinces, Yunnan has the highest number of reported HIV infections in China whereas Fujian is one of the provinces reporting the lowest HIV prevalence rate in China. With the trial implemented in Yunnan and Fujian Provinces simultaneously, we will examine the program's efficacy in two provinces that vary dramatically in HIV prevalence and infection routes. We propose to include two provinces that represent China as a whole, due to the varied HIV rates and infection routes in diverse regions; thus allowing us to disentangle the relations among HIV-related stigma, fear of infection, and HIV prevalence.

Specific Aim 1: To examine whether providers in the intervention hospitals, compared to providers in the standard care condition, will demonstrate positive attitudinal outcomes, including an increase in comfort in working with PLH and a decrease in unrealistic fear of infection at work, prejudicial attitudes, and support of coercive policies.

Specific Aim 2: To examine whether providers in the intervention hospitals, compared to providers in the standard care condition, will demonstrate more positive behavioral outcomes, including an increase in adherence to universal precaution, routine treatment and referrals, confidentiality protection, diffusion of positive messages with co-workers, and a decrease in critical incidents.

Specific Aim 3: To explore whether patients in the intervention hospitals, compared to patients at hospitals in the standard care condition, will report a decreased level of perceived unfair treatment and increased service satisfaction, service utilization, and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Service providers: 18 years and older, who work at the county hospital that is participating in the study, including doctors, nurses and lab technicians, and who provide informed consent.
* Hospital administrators: 18 years and older, who work at the county hospital that is participating in the study as administrators, and who provide informed consent.
* Patients: Age 18 and older, who receive treatment from STD, obstetrics/gynecology or HIV care department at the participating hospital, and who provide informed consent.

Exclusion Criteria:

* Those who cannot give informed consent (e.g., intoxicated)
* Those who have a permanent disability (e.g., deaf, serious mental illness, mental retardation).
* Anyone who does not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5400 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
HIV related stigma | 6-month and 12-month follow-up
Patient satisfaction | 6-mont and 12-month follow-up

SECONDARY OUTCOMES:
Universal precaution | 6-month and 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, PhD, Principal Investigator — UCLA Semel Institute, Center for Community Health
Locations (1):
- UCLA Semel Institute-Center for Community Health, Los Angeles, California, United States

REFERENCES:
- [Result] Li L, Liang LJ, Wu Z, Lin C, Guan J. Assessing outcomes of a stigma-reduction intervention with venue-based analysis. Soc Psychiatry Psychiatr Epidemiol. 2014 Jun;49(6):991-9. doi: 10.1007/s00127-013-0808-6. Epub 2013 Dec 28. PMID 24374721
- [Result] Li L, Wu Z, Liang LJ, Lin C, Guan J, Jia M, Rou K, Yan Z. Reducing HIV-related stigma in health care settings: a randomized controlled trial in China. Am J Public Health. 2013 Feb;103(2):286-92. doi: 10.2105/AJPH.2012.300854. Epub 2012 Dec 13. PMID 23237175